CLINICAL TRIAL: NCT03075969
Title: An International Field Study for the Reliability and Validity of the Phase IV EORTC Quality of Life Module for Patients With Chronic Myeloid Leukemia (EORTC QLQ-CML24)
Brief Title: Phase IV EORTC Quality of Life Module for Patients With Chronic Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QoL-CML 0916
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic myeloid leukemia; quality of life
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to test the scale structure, reliability, validity and responsiveness to change of the QLQ-CML24 in conjuction with the QLQ-C30 for patients diagnosed with CML, and to investigate longitudinal relationship between satisfaction with information provision and QoL outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age.
* Patient with confirmed diagnosis of Philadelphia chromosome positive and/or BCR-ABL positive chronic myeloid leukemia (CML).
* Written informed consent.
* Patients enrolled in investigational drug-trials or other type of clinical trials are also eligible.

Exclusion Criteria:

* Patients with a psychiatric condition or major cognitive impairment (as evaluated by their treating physician) that would hinder completion of self-reported health-related QoL questionnaires.
* Patients who are unable to speak and read the language of the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be composed of four different groups of patients in order to achieve the purposes of this field-testing.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-03-16 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to test the scale structure, reliability, validity and responsiveness to change of the QLQ-CML24 in conjunction with the QLQ-C30 for patients diagnosed with CML. | 18 months from enrollment

SECONDARY OUTCOMES:
The secondary objective is to investigate longitudinal relationship between satisfaction with information provision (outcome measure: EORTC INFO-25) and QoL outcomes (outcome measures: EORTC QLQ-C30 and QLQ-CML24). | 18 months from enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Efficace, PhD, Study Chair — GIMEMA Foundation
Locations (32):
- Winship Cancer Institute of Emory University, Emory, Georgia, United States
- Innsbruck Medical University, Innsbruck, Austria
- Complexo Hospital de Clinicas da Universidade Federal do Parana, Paranã, Brazil
- Guangdong Medical University, Guangdong, China
- Universität Heidelberg, Heidelberg, Germany
- Baghdad Teaching Hospital, Baghdad, Iraq
- Italy (24):
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
  - Azienda Ospedaliero-Universitaria Policlinico Consorziale, Bari
  - Department of Oncology and Hematology, O.U. of Hematology, S. Orsola-Malpighi University Hospital, Bologna, Bologna
  - Sezione di Ematologia e Trapianti Spedali Civili, Brescia
  - CTMO - Ematologia - Ospedale Binaghi, Cagliari
  - Divisione clinicizzata di Ematologia - Dipartimento di Scienze Mediche - Osp. Ferrarotto, Catania
  - Clinica Ematologica - Dipartimento di Medicina Interna - IRCCS San Martino - IST, Genova
  - Lecce ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - U.O. Ematologia 1 - Centro Trapianti di Midollo - Ospedale Maggiore Milano, Milan
  - Divisione di Ematologia - Dip. Di Medicina Clinica e Sperimentale & BRMA - Università Piemonte Orientale "Amedeo Avogato", Novara
  - Azienda Ospedaliera Universitaria - Policlinico Paolo Giaccone, Palermo
  - U.O.C. di Ematologia e CTMO Az. Ospedaliero Universitaria Parma, Parma
  - Div. di Ematologia IRCCS Policlinico S. Matteo, Pavia
  - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Clinica di Ematologia - Policlinico Umberto I- Università degli Studi "Sapienza", Roma
  - Divisione di Ematologia - Ospedale S.Eugenio, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - U.O. di Ematologia - Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - AOU Sassari, Sassari
  - U.O di Ematologia d. U. - Azienda Ospedaliera Universitaria Integrata Verona, Verona
  - Ospedale San Bortolo, Vicenza
- UCSI University, Faculty of Pharmaceutical Sciences, Kuala Lumpur, Malaysia
- Eindhoven and Tilburg University, Eindhoven, Netherlands